CLINICAL TRIAL: NCT01249677
Title: Chronic Reduction of Fasting Gylcaemia With Insulin Glargine Improves First and Second Phase Insulin Secretion in Patients With Type 2 Diabetes
Brief Title: Chronic Reduction of Fasting Glycaemia With Insulin Glargine Improves First and Second Phase Insulin Secretion in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Prof. Dr. Wolfgang E. Schmidt; Director Department of Medicine I, University Hospital; Ruhr-University Bochum; Gudrunstr. 56; 44791 Bochum; Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08- BO-LSBE
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2008-10

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; first phase insulin secretion; beta-cell rest; basal insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- insulin glargine (Experimental): patients with type 2 diabetes on previous therapy with metformin were examined before and after eight weeks of treatment with insulin glargin, aimed to normalize fasting plasma glycaemia
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin glargine — 14 patients with type 2 diabetes on previous metformin therapy were treated with insulin glargine, aimed to normalize fasting glycaemia.
  Other Names: Lantus

SUMMARY:
Glucose-induced insulin secretion is often diminished in hyperglycaemic patients with type 2 diabetes. The investigators examined, whether chronic basal insulin treatment with insulin glargine lead to improvements in glucose-induced insulin secretion.

DETAILED DESCRIPTION:
14 patients with type 2 diabetes on previous metformin therapy were examined before and after eight weeks of treatment with insulin glargine, aimed to normalize fasting glycaemia. Intravenous glucose tolerance tests were performed with and without previous adjustment of fasting glucose levels by means of a 3-hour intravenous insulin infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 75 years, inclusive
2. BMI-range 27-50 kg/m²
3. patients with type 2 diabetes presenting with fasting hyperglycaemia (>126mg/dl) on metformin treatment

Exclusion Criteria:

1.Pre-existing insulin therapy, treatment with sulphonylureas, glitazones, 2.glinides, DPP-4-inhibitors or exenatide 3.patients with type 1 diabetes 4.Patients are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.

5. Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures include sterilisation, hormonal intrauterine devices, oral contraceptives, sexual abstinence or vasectomised partner). A male subject who is sexually active and has not been surgically sterilised must be informed that he must either use a condom during intercourse, ensure that his partner practices contraception, or he must refrain from sexual intercourse during the trial and until 1 month after completion of the trial. This is to prevent the possibility of a pregnancy from spermatocytes that can potentially be damaged by trial medication. It is strongly recommended that the female partners use a highly effective contraception (Pearl Index < 1%).

6. Patients have participated in an interventional medical, surgical, or pharmaceutical study (a study in which an experimental, drug, medical, or surgical treatment was given) within 30 days prior to screening. This criterion includes drugs that have not received regulatory approval for any indication at the time of study entry.

7. Patients have alcohol consumption (>20 g daily for males and >10 g daily for females) 8. Patients have alanine aminotransaminase (ALT) greater than ten times the upper limit of the reference range.

9.Patients are undergoing therapy for a malignancy, other than basal cell or squamous cell skin cancer.

10. Patients have cardiac disease that is Class III or IV, according to the New York Heart Association criteria.

11. Patients have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine >1.8 mg/dL for males and greater than or equal to >1.5 mg/dL for females. 12.Patients have known hemoglobinopathy or chronic anemia 13.Patients are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks immediately prior to screening.

14. Patients have any other condition (including known drug or alcohol abuse or psychiatric disorder) that precludes them from following and completing the protocol, in the opinion of the investigator.

15. Patients fail to satisfy the investigator of suitability to participate for any other reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Improvements in first and second phase insulin secretion | 8 weeks
  Improvements in first and second phase insulin secretion after bedtime administration of insulin glargin, titrated to reach normal (90-100 mg/dl) fasting glucose levels

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine I; University Hospital St. Josef Hospital, Bochum, Germany

REFERENCES:
- [Derived] Pennartz C, Schenker N, Menge BA, Schmidt WE, Nauck MA, Meier JJ. Chronic reduction of fasting glycemia with insulin glargine improves first- and second-phase insulin secretion in patients with type 2 diabetes. Diabetes Care. 2011 Sep;34(9):2048-53. doi: 10.2337/dc11-0471. Epub 2011 Jul 20. PMID 21775756